CLINICAL TRIAL: NCT03784794
Title: ROTEM Guided and Hemostatic Drugs Algorithms vs Standard Coagulation Test and Hemocomponent for Massive Obstetric Hemorrhage
Brief Title: Patient Blood Management for Massive Obstetric Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Angel Augusto Perez Calatayud (Other)
Collaborators: Grupo Mexicano para el Estudio de la Medicina Intensiva (Other)
Responsible Party: Sponsor-Investigator, Angel Augusto Perez Calatayud, Head Intensive Care Unit Hospital de Especialidades del Niño y la Mujer Dr Felipe Nuñez Lara, Grupo Mexicano para el Estudio de la Medicina Intensiva
Organization: Grupo Mexicano para el Estudio de la Medicina Intensiva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 099/21012018/MEDCRITICAHENM
Record Dates: First submitted 2018-12-14; First posted 2018-12-24 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Post Partum Hemorrhage; Fibrinogenolysis; Hemorrhage; Fibrinogen; Deficiency, Acquired; Massive Hemorrhage; Transfusion Related Complication
Keywords: Post Partum Hemorrhage; Massive tranfusion; Thromboelastometry
MeSH Terms: conditions — Postpartum Hemorrhage; Disseminated Intravascular Coagulation | interventions — Thrombelastography; Blood Coagulation Tests; Fibrinogen; prothrombin complex concentrates; Platelet Count; Erythrocyte Count

STUDY DESIGN:
Intervention Model Description: Group A Fibrinogen Concentrate, Protrombin Complex Concentrate, trhromboelastometry guided Group B Cryoprecipitates, fresh frozen plasma, standard coagulation lab test
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thromboelastometry (Experimental): Decision to treat will be guided with thromboelastometry results, for fribrinogen deficiency the investigators will treat with fibrinogen concentrate (human), for correction of factor deficiency Prothrombin Complex Concentrates, Platelets with the use of platelets and Red Blood Cells for correcting hemoglobin levels
  Interventions: Diagnostic Test: Thromboelastometry; Drug: Fibrinogen Concentrate Human; Drug: Prothrombin Complex Concentrates; Other: Platelets; Other: Red Blood Cells
- STANDARD COAGULATION TEST ALGORITHM (Active Comparator): Decision to treat will be guided by standard cogulation lab test (Thrombine time, Active Thromboplastine time, Clauss fibrinogen, platelets count etc) for fribrinogen deficiency the investigators will treat with cryoprecipitates, for correction of factor deficiency fresh frozen plasma, Platelets with the use of platelets and Red Blood Cells for correcting hemoglobin levels
  Interventions: Diagnostic Test: Standard Coagulation Test; Other: Platelets; Other: Red Blood Cells; Other: Fresh Frozen Plasma; Other: cryoprecipitates

INTERVENTIONS:
Diagnostic Test: Thromboelastometry — devices generate output by transducing changes in the viscoelastic strength of a small sample of clotting blood (300 µl) to which a constant rotational force is applied. These point of care devices allow visual assessment of blood coagulation from clot formation, through propagation, and stabilization, until clot dissolution. Computer analysis of the output allows sophisticated clot formation/dissolution kinetics and clot strength data to be generated
  Other Names: ROTEM
  Arms: Thromboelastometry
Diagnostic Test: Standard Coagulation Test — coagulation tests, such as the prothrombin time (PT), activated partial thromboplastin time (aPTT), and thrombin time (TT), to assess blood clotting function in patients. Clauss Fibrinogen.
  Other Names: blood coagulation test
  Arms: STANDARD COAGULATION TEST ALGORITHM
Drug: Fibrinogen Concentrate Human — To treat acquired fribinogen deficiency investigators will treat with the following doses FIBTEM A5 = 9-11 MM a 2 G FIBRINOGEN CONC. (25 MG/KG); FIBTEM A5 = 4-8 MM a 4 G FIBRINOGEN CONC. (50 MG/KG); FIBTEM A5 < 4 MM a 6 G FIBRINOGEN CONC. (75 MG/KG)
  Other Names: Chlotafact
  Arms: Thromboelastometry
Drug: Prothrombin Complex Concentrates — to treat acquired factor deficiency investigators will treat as follows PROTROMBIN COMPLEX CONCENTRATE EXTEM CT > 80 SEC AND FIBTEM A5 ≥ 8 MM 4F-PCC 20 IU/KG (F II, VII, IX and X) GOAL: EXTEM CT ≤ 80 SEC
  Other Names: Confidex
  Arms: Thromboelastometry
Other: Platelets — PLATELETS EXTEM A5 < 40 MM AND FIBTEM A5 ≥ 12 MM EXTEM A5 < 40 MM → 1 PLATELET POOL OR APHERESIS; EXTEM A5 < 30 MM → 2 PLATELET POOL OR APHERESIS GOAL: EXTEM A5: 40-50 MM or PLATELET COUNT < 100/µL PLT < 100/µL → 1 PLATELET POOL OR APHERESIS; PLT > 50/µL → 2 PLATELET POOL OR APHERESIS GOAL: PLT COUNT > 100/µL
Other: Red Blood Cells — Transfuce Red Blood Cells if Hemoglobine levels < 7 G/DL;
  1 unit of FFP for every unit of RBC Transfused GOAL: Hb > 7.5 G/DL
  Other Names: RBC
Other: Fresh Frozen Plasma — FRESH FROZEN PLASMA TP AND/OR TTP PATHOLOGICAL INR, 2.0-4.0 → FFP 20 ML/KG GOAL: TP AND TTP NORMAL AND INR < 2.0
  Arms: STANDARD COAGULATION TEST ALGORITHM
Other: cryoprecipitates — FIBRINOGEN (CLAUSS) < 250 MG/DL FIB 200-250 MG/DL → CRYOS, PACK OF 10 (25 MG/KG); FIB 100-200 MG/DL → CRYOS, PACK OF 20 (50 MG/KG); FIB < 100 MG/DL → CRYOS, PACK OF 30 (75 MG/KG) GOAL: FIB > 250 MG/DL
  Arms: STANDARD COAGULATION TEST ALGORITHM

SUMMARY:
Obstetric Hemorrhage continues to be the first cause of maternal morbidity and mortality around the world especially in middle to low income countriesThe blood components are high value resources; however, its use has been shown to be a risk factor of known complications. The aim of the study is to compare two algorithms of coagulation management in massive obstetric hemorrhage Methods A randomized prospective trial single center two arms study in patients with severe obstetric hemorrhage (PPH > 1000) 2 different transfusion protocols one guided by thromboelastometry and hemostatic drugs (protrombine complex concentrate and fibrinogen concentrate) and the second guided by standard coagulation test and hemocomponents. Sample is calculated to known variance, Analyses are intention-to-treat without imputation, with outcomes will be performed between groups using mixed-effects two level regression models. For binary outcomes, a logistic model will be used and results presented as adjusted odds ratios (ORs) alongside 95% confidence intervals (CIs). Count data will be analysed using Poisson multilevel or negative binomial models.

Primary Outcome Parameter:

Compare between the two protocols:

Number of allogeneic blood products transfused intra-op, within 24h after screening and in-hospital (RBC, Platelets and FFP; separate and overall)

Secondary Outcome Parameter:

Analysis of mortality, lenth of stay admission to the ICU, hysterectomy surgical reintervencion, Transfuse associated circulatory overload, Transfusion associated Acute lung injury, health associated infection will be measured as secondary outcome.

DETAILED DESCRIPTION:
Introduction Obstetric Hemorrhage continues to be the first cause of maternal morbidity and mortality around the world especially in middle to low income countries. Copying trauma transfusion therapies now a days algorithms have been developing for 2.1.1 transfusion in massive obstetric hemorrhage. Blood products, play an essential role in the management of these patients, either during resuscitation or definitive treatment. Early transfusion, defined as that required in the first 24 hours after admission, it is required in about 5% that enters the hospital and about 3% comes to require massive transfusion. The blood components are high value resources; however, its use has been shown to be a risk factor for infectious transfusion related immunomodulation, and noninfectious complications (TRALI, TACO), development of systemic inflammatory response, multiple organ failure and death. A liberal transfusion policy can further introduce the risk of a patient who is already committed.

Patient blood management is an evidence-based, multidisciplinary approach to optimizing the care of patients who might need transfusion. PBM encompasses all aspects of patient evaluation and clinical management surrounding the transfusion decision-making process, including the application of appropriate indications, as well as minimization of blood loss and optimization of patient red cell mass.

The aim of the study is to compare two algorithms of coagulation management in massive obstetric hemorrhage Methods A randomized prospective trial single center two arms study in patients with severe obstetric hemorrhage (PPH > 1000) 2 different transfusion protocols one guided by thromboelastometry and hemostatic drugs (protrombine complex concentrate and fibrinogen concentrate) and the second guided by standard coagulation test and hemocomponents.

Randomization for the patients will be made for every obstetric patient that enters the obstetric ward for attention of partum, and will be asked to sign consent, and the patients will be selected for each group of the study. Only does that have severe PPH will be entering the protocol with the algorithm for management previously selected. Demographic caracteristics will include Ethnicity, Body weight (KG), body height (CM) and BMI at hospital admission, Previous deliveries, Previous Caesarean section, Pre-eclampsia during pregnancy, History of obstetric hemorrhage, History of other kind of hemorrhage, Onset of labor (spontaneous, induced, no labor) Multiple gestation (singleton, twins, triplet) Reported cause of obstetric hemorrhage (placenta previa, placenta accreta, placenta abruption, retained placenta, uterine atony, trauma, surgical bleeding Mode of delivery (spontaneous vaginal, instrumental vaginal , elective Caesarean section, non-elective Caesarean section) Baseline Hb, Hct, Plt count, Fibrinogen (Clauss), PT/INR, PTT (at hospital admission) Estimated blood loss at study entry (ML).

Treatment algorithms are evidence based and the management of coagulopathy is based on treat first what kills fist (ATLS proposal)

Group A:

THROMBOELASTOMETRY-GUIDED ALGORITHM FIBRINOGEN CONCENTRATE FIBTEM A5 < 12 MM AND EXTEM A5 < 40 MM FIBTEM A5 = 9-11 MM → 2 G FIBRINOGEN CONC. (25 MG/KG); FIBTEM A5 = 4-8 MM → 4 G FIBRINOGEN CONC. (50 MG/KG); FIBTEM A5 < 4 MM → 6 G FIBRINOGEN CONC. (75 MG/KG) GOAL: FIBTEM A5: 12-16 MM PLATELETS EXTEM A5 < 40 MM AND FIBTEM A5 ≥ 12 MM EXTEM A5 < 40 MM → 1 PLATELET POOL OR APHERESIS; EXTEM A5 < 30 MM → 2 PLATELET POOL OR APHERESIS GOAL: EXTEM A5: 40-50 MM PROTROMBIN COMPLEX CONCENTRATE EXTEM CT > 80 SEC AND FIBTEM A5 ≥ 8 MM 4F-PCC 20 IU/KG (F II, VII, IX and X) GOAL: EXTEM CT ≤ 80 SEC NO INTERVENTION FIBTEM A5 ≥ 12 MM AND EXTEM A5 ≥ 40 MM AND EXTEM CT > 80 SEC NO FIBRINOGEN, CRYO, PLATELETS, 4-PCC, FFP; TRANSFUSE RBC IF Hb < 7 G/DL GOAL: Hb > 7.5 G/DL

Group B RATIO / STANDRAD LAB TEST-GUIDED ALGORITHM CRYOPRECIPITATE FIBRINOGEN (CLAUSS) < 250 MG/DL FIB 200-250 MG/DL → CRYOS, PACK OF 10 (25 MG/KG); FIB 100-200 MG/DL → CRYOS, PACK OF 20 (50 MG/KG); FIB < 100 MG/DL → CRYOS, PACK OF 30 (75 MG/KG) GOAL: FIB > 250 MG/DL PLATELETS PLATELET COUNT < 100/µL PLT < 100/µL → 1 PLATELET POOL OR APHERESIS; PLT > 50/µL → 2 PLATELET POOL OR APHERESIS GOAL: PLT COUNT > 100/µL FRESH FROZEN PLASMA TP AND/OR TTP PATHOLOGICAL INR, 2.0-4.0 → FFP 20 ML/KG GOAL: TP AND TTP NORMAL AND INR < 2.0 NO LAB RESULTS AVAILABLE TRANSFUSE RED BLOOD CELLS IF Hb < 7 G/DL; GIVE 1 UNIT FFP EVERY 2 UNITS OF RBC TRANSFUSED GOAL: Hb > 7.5 G/DL Statistical analysis Sample is calculated to known variance. The investigators calculated that 100 women will be needed to provide 80% power at the two-sided 5% level to detect a difference of total allogeneic units between groups. With a total of 100 patients 50 in each arm, with a first revision of results after recruiting 50 patients (25 in each arm). Analyses are intention-to-treat without imputation, with outcomes will be performed between groups using mixed-effects two level regression models. For binary outcomes, a logistic model will be used and results presented as adjusted odds ratios (ORs) alongside 95% confidence intervals (CIs). For continuous outcomes, a linear regression model will be performed and results presented as difference in adjusted means (arm A vs arm B) alongside 95% CIs. Count data will be analysed using Poisson multilevel or negative binomial models if over-dispersion is evident and presented as incident rate ratios (IRRs).

Objectives

Primary Outcome Parameter:

Compare between the two protocols:

Number of allogeneic blood products transfused intra-op, within 24h after screening and in-hospital (RBC, Platelets and FFP; separate and overall)

Secondary Outcome Parameter:

Compare between the two arms Number of packs of Cryo (pack of 5 ~ 1 G Fibrinogen), Fibrinogen Concentrate (G), and PCC (500 UI) administered intra-op, within 24h after screening and in-hospital Incidence ≥ 5 U RBC transfused (first 24h after screening) Incidence ≥ 10 U RBC transfused (first 24h after screening) Incidence of RBC, Platelets, FFP, Cryo, Fibrinogen Concentrate, and PCC transfusion/administration (intra-op, first 24h and in-hospital) Total volume of blood products and coagulation factor concentrates transfused/administered (intra-op, first 24h and in-hospital) Infusion: Crystalloid (ML) and Colloids (Type; ML) intra-op and within 24h after screening Overall estimated blood loss (EBL, ML) Time to bleeding control (time from study entry to last hemostatic intervention/transfusion) Incidence of coagulopathy (detected by thromboelastometry or standard coagulation laboratory tests) Incidence of hysterectomy Incidence of re-surgery Incidence of TACO Incidence of TRALI Incidence of surgical site infection or sepsis Incidence of ICU admission Length of stay (LOS) at ICU and hospital In-hospital mortality First post-op Hb, Hct, Plt count, Fibrinogen (Clauss), PT, INR, PTT (recovery room or ICU) Last Hb, Hct, Plt count, Fibrinogen (Clauss), PT, INR, PTT before discharge from hospital Total acquisition costs of allogeneic blood products and coagulation factor concentrates HYPOTHESIS. The algorithm guided by ROTEM plus the use of hemostatic drugs, are more efficient for the reversion of coagulopathy due to obstetric hemorrhage, than the standard treatment group, decrases the risk of development known complications, decreases the need of blood transfusions, decreases morbidity and mortality associated to PPH, length of stay, admissions to the intensive care unit and days of mechanical ventilation. Without a significant increase in costs.

RELEVANCE AND EXPECTATIONS To offer a safe alternative in the treatment of severe obstetric hemorrhage, which reduces the risk of transfusion associated complications,

ELIGIBILITY:
Inclusion Criteria:

Patients with severe obstetric hemorrhage of any cause

Exclusion Criteria:

obstetric hemorrhage patients derived from other hospitals Patients with less than 1000 ml of estimated blood loss those who do not want to participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — all female patients with severe obstetric hemorrhage (more than 1000 ml of estimated blood loss)
Enrollment: 100 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Number of Blood products transfused | 24 hrs
  Number of allogeneic blood products transfused intra-op, within 24h after screening and in-hospital (RBC, Platelets and FFP; separate and overall)

SECONDARY OUTCOMES:
Number of hemocomponents or fibrinogen concentrates needed to treat hypofibrinogenemia | day 0 to day 15
  Number of packs of Cryo (pack of 5 ~ 1 G Fibrinogen), Fibrinogen Concentrate (G), and PCC (500 UI) administered intra-operating
Incidence of Red Blood Cells transfusion (RBC) | day 0 to day 15
  Incidence ≥ 5 U RBC transfused
Incidence of Massive Red Blood Cells transfusion (RBC) | day 0 to day 15
  Incidence ≥ 10 U RBC transfused (first 24h after screening)
estimated blood loss | day 0 to day 15
  Overall estimated blood loss (EBL, ML)
Time to bleeding control | 24 hrs
  time from study entry to last hemostatic intervention/transfusion
Incidence of coagulopathy | day 0 to day 15
  detected by thromboelastometry or standard coagulation laboratory tests
Incidence of hysterectomy | day 0 to day 15
  number of obstetric hysterectomy for bleeding control
Incidence of re-surgery | day 0 to day 15
  number of procedures necessary for bleeding control
Incidence of Transfused associated circulatory overload | day 0 to day 15
  number of patients with transfused associated circulatory overload
Incidence of surgical site infection or sepsis | day 0 to day 15
  number of patients that developed health care related infections or sepsis
Incidence of ICU admission | day 0 to day 15
  number of patients that require admission to the ICU for complications related to hipovolemic shock
In-hospital mortality | day 0 to day 15
  number of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Angel Augusto Perez Calatayud, M.D., Principal Investigator — Head Obstetric ICU
Locations (1):
- Hospital de Especialidades Del Niño Y La Mujer, Querétaro City, Querétaro, Mexico

IPD SHARING:
Plan to Share IPD: Yes
no plan for sharing data has been made
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after recruiting 50% of the participants and it will be available always
Access Criteria: open

REFERENCES:
- [Background] Mallaiah S, Barclay P, Harrod I, Chevannes C, Bhalla A. Introduction of an algorithm for ROTEM-guided fibrinogen concentrate administration in major obstetric haemorrhage. Anaesthesia. 2015 Feb;70(2):166-75. doi: 10.1111/anae.12859. Epub 2014 Oct 7. PMID 25289791
- [Background] Mallaiah S, Chevannes C, McNamara H, Barclay P. A reply. Anaesthesia. 2015 Jun;70(6):760-1. doi: 10.1111/anae.13128. No abstract available. PMID 25959192
- [Background] Collins PW, Cannings-John R, Bruynseels D, Mallaiah S, Dick J, Elton C, Weeks AD, Sanders J, Aawar N, Townson J, Hood K, Hall JE, Collis RE. Viscoelastometric-guided early fibrinogen concentrate replacement during postpartum haemorrhage: OBS2, a double-blind randomized controlled trial. Br J Anaesth. 2017 Sep 1;119(3):411-421. doi: 10.1093/bja/aex181. PMID 28969312
- [Background] Wikkelso AJ, Edwards HM, Afshari A, Stensballe J, Langhoff-Roos J, Albrechtsen C, Ekelund K, Hanke G, Secher EL, Sharif HF, Pedersen LM, Troelstrup A, Lauenborg J, Mitchell AU, Fuhrmann L, Svare J, Madsen MG, Bodker B, Moller AM; FIB-PPH trial group. Pre-emptive treatment with fibrinogen concentrate for postpartum haemorrhage: randomized controlled trial. Br J Anaesth. 2015 Apr;114(4):623-33. doi: 10.1093/bja/aeu444. Epub 2015 Jan 13. PMID 25586727
- [Background] Snegovskikh D, Souza D, Walton Z, Dai F, Rachler R, Garay A, Snegovskikh VV, Braveman FR, Norwitz ER. Point-of-care viscoelastic testing improves the outcome of pregnancies complicated by severe postpartum hemorrhage. J Clin Anesth. 2018 Feb;44:50-56. doi: 10.1016/j.jclinane.2017.10.003. Epub 2017 Nov 7. PMID 29121548
- [Background] Olde Engberink RH, Kuiper GJ, Wetzels RJ, Nelemans PJ, Lance MD, Beckers EA, Henskens YM. Rapid and correct prediction of thrombocytopenia and hypofibrinogenemia with rotational thromboelastometry in cardiac surgery. J Cardiothorac Vasc Anesth. 2014 Apr;28(2):210-6. doi: 10.1053/j.jvca.2013.12.004. PMID 24630470
- [Background] Song JG, Jeong SM, Jun IG, Lee HM, Hwang GS. Five-minute parameter of thromboelastometry is sufficient to detect thrombocytopenia and hypofibrinogenaemia in patients undergoing liver transplantation. Br J Anaesth. 2014 Feb;112(2):290-7. doi: 10.1093/bja/aet325. Epub 2013 Sep 24. PMID 24065728
- [Background] Collins PW, Lilley G, Bruynseels D, Laurent DB, Cannings-John R, Precious E, Hamlyn V, Sanders J, Alikhan R, Rayment R, Rees A, Kaye A, Hall JE, Paranjothy S, Weeks A, Collis RE. Fibrin-based clot formation as an early and rapid biomarker for progression of postpartum hemorrhage: a prospective study. Blood. 2014 Sep 11;124(11):1727-36. doi: 10.1182/blood-2014-04-567891. Epub 2014 Jul 14. PMID 25024304
- [Background] Hagemo JS, Christiaans SC, Stanworth SJ, Brohi K, Johansson PI, Goslings JC, Naess PA, Gaarder C. Detection of acute traumatic coagulopathy and massive transfusion requirements by means of rotational thromboelastometry: an international prospective validation study. Crit Care. 2015 Mar 23;19(1):97. doi: 10.1186/s13054-015-0823-y. PMID 25888032
- [Background] Baksaas-Aasen K, Van Dieren S, Balvers K, Juffermans NP, Naess PA, Rourke C, Eaglestone S, Ostrowski SR, Stensballe J, Stanworth S, Maegele M, Goslings JC, Johansson PI, Brohi K, Gaarder C; TACTIC/INTRN collaborators. Data-driven Development of ROTEM and TEG Algorithms for the Management of Trauma Hemorrhage: A Prospective Observational Multicenter Study. Ann Surg. 2019 Dec;270(6):1178-1185. doi: 10.1097/SLA.0000000000002825. PMID 29794847
- [Background] Mace H, Lightfoot N, McCluskey S, Selby R, Roy D, Timoumi T, Karkouti K. Validity of Thromboelastometry for Rapid Assessment of Fibrinogen Levels in Heparinized Samples During Cardiac Surgery: A Retrospective, Single-center, Observational Study. J Cardiothorac Vasc Anesth. 2016 Jan;30(1):90-5. doi: 10.1053/j.jvca.2015.04.030. Epub 2015 May 5. PMID 26296822
- [Result] Perez-Calatayud AA, Briones-Garduno JC, Rojas-Arellano ML. [Use of thromboelastography and thromboelastometry for the rational and opportune transfusion of hemoderivatives in obstetric hemorrhage]. Ginecol Obstet Mex. 2015 Sep;83(9):569-77. Spanish. PMID 26591047